CLINICAL TRIAL: NCT03056638
Title: Phase III Randomized Trial Comparing Short Course Androgen Deprivation Therapy and Ultra-Hypofractionated SBRT Versus SBRT Alone For Intermediate Prostate Cancer
Brief Title: Trial of ADT and SBRT Versus SBRT for Intermediate Prostate Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to low accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Ferring Pharmaceuticals (Industry); University of Texas Southwestern Medical Center (Other); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1686
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
Keywords: Androgen Deprivation Therapy; Ultra-Hypofractionated SBRT; 16-1686
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Eligible patients with intermediate risk disease will be randomized to ADT with SBRT versus SBRT alone. PSA and testosterone testing every 6 months, Biopsy 24-30 months after SBRT
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Degarelix in conjunction with stereotactic body radiosurgery (Experimental): Degarelix monthly for 6 months SBRT 8 Gy x 5
  Interventions: Drug: Degarelix; Radiation: stereotactic body radiosurgery (SBRT)
- stereotactic body radiosurgery (SBRT) (Experimental): SBRT 8 Gy x 5
  Interventions: Radiation: stereotactic body radiosurgery (SBRT)

INTERVENTIONS:
Drug: Degarelix — Degarelix monthly for 6 months
  Arms: Degarelix in conjunction with stereotactic body radiosurgery
Radiation: stereotactic body radiosurgery (SBRT) — SBRT 8 Gy x 5

SUMMARY:
Stereotactic body radiation therapy (SBRT) is a very precise form of radiation therapy that allows the physician to deliver more radiation dose in a single session. Because of this, the number of radiation sessions can be reduced from the typical 45-48 sessions, as in conventional daily session radiation, to 5 sessions given every other day over a week and a half. Giving the radiation at a higher dose during each treatment may be more effective in killing the prostate cancer cells than the standard way of using external radiation therapy where a small amount of radiation is given over many sessions.

Androgen Deprivation Therapy (ADT) or hormonal therapy is one of the methods to treat intermediate risk prostate cancer. This therapy works by reducing the level of testosterone and stopping them from affecting your cancer. The ADT used in this study is known as Degarelix. Degarelix is an approved medication that reduces the body's production of testosterone; this medication is usually given to all men with intermediate risk prostate cancer getting external radiation.

This study is a randomized study to find out whether combining stereotactic (also known as precision) radiation to the prostate cancer combined with a short course of Degarelix will result in a greater likelihood of killing the cancer in the prostate compared to stereotactic radiation therapy given alone. It has been shown that the combination of radiation with medications that interfere with testosterone production and its effects makes prostate cancer cells more sensitive to the radiation.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven intermediate risk prostate cancer, which includes patients with any one of the following variables:
* Gleason 7 disease
* PSA 10-20 ng/ml
* Clinical T2b-T2c disease Note: Patients who only have radiographic evidence of T3 disease (i.e. extracapsular extension, or seminal vesical invasion radiographically) will not be excluded.
* Serum testosterone ≥ 240 ng/dL determined within 2 months prior to enrollment
* At least 4 weeks must have elapsed from major surgery
* KPS ≥ 80%
* Prostate size as determined on MRI to be < 90 cc. Prostate size can be determined on CT scan if MRI is not available.
* 18 years of age or older
* IPSS ≤ 20
* Patient must be available for follow-up. After 2 years of follow-up following post-treatment biopsy, telephone-based follow-up will be acceptable
* Laboratory test findings within 8 weeks of randomization:

  * Adequate hepatic function with serum bilirubin ≤ 1.5 times the upper institutional limits of normal (ULN), ALT and AST ≤ 2.5 x ULN. Patients with a history of Gilbert's syndrome may be enrolled if the total bilirubin is < 3 mg/dL with a predominance of indirect bilirubin
  * Adequate renal function with serum creatinine ≤ 1.5 x ULN
  * Adequate hematologic function with absolute neutrophil counts ≥ 1,500 cell/mm3 and platelets ≥ 100,000 cells/mm3 and hemoglobin value ≥ 9 g/dL (Note: patients whose anemia has been corrected to a hemoglobin value ≥ 9 g/dL with blood transfusions are allowed)

Exclusion Criteria:

* CT or MRI evidence of metastatic disease to the bone.
* Patients with one or more positive lymph nodes considered suspicious as determined by clinical assessment on MRI or CT
* Prior treatment for prostate cancer, including history of chemotherapy, hormonal therapy within 30 days of enrollment or surgery for prostate cancer (except for prior TURP or greenlight PVP which would be allowed)
* History of another malignancy within the previous 3 years except for the following: adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, currently in complete remission, or any other cancer that has been in complete remission for at least 3 years
* Patients with Crohn's disease or ulcerative colitis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — prostate cancer
Enrollment: 56 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zelefsky, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Baptist Alliance MCI, Miami, Florida
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Degarelix in Conjunction With Stereotactic Body Radiosurgery | Stereotactic Body Radiosurgery (SBRT)
Started | 27 | 29
Completed | 26 | 29
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix in Conjunction With Stereotactic Body Radiosurgery | Stereotactic Body Radiosurgery (SBRT) | Total
Number analyzed (Participants) | 27 | 29 | 56
Age, Continuous [Median (Full Range); unit: years] | 68 [54 to 79] | 70 [55 to 79] | 68 [54 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 27 | 29 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 24 | 26 | 50
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 19 | 19 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 29 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Positive Biopsy
Description: compare 2-year biopsy positivity rate of intermediate risk prostate cancer patients treated with SBRT + short course ADT versus SBRT alone.
Time Frame: 2 years
Population: N/A - data were not collected
Arm/Group | Degarelix in Conjunction With Stereotactic Body Radiosurgery | Stereotactic Body Radiosurgery (SBRT)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Degarelix in Conjunction With Stereotactic Body Radiosurgery | Stereotactic Body Radiosurgery (SBRT)
All-Cause Mortality (participants affected / at risk) | 1/27 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/27 | 0/29
Other Adverse Events (participants affected / at risk) | 2/27 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Degarelix in Conjunction With Stereotactic Body Radiosurgery (N=27) | Stereotactic Body Radiosurgery (SBRT) (N=29)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Degarelix in Conjunction With Stereotactic Body Radiosurgery (N=27) | Stereotactic Body Radiosurgery (SBRT) (N=29)
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT03056638/Prot_SAP_000.pdf